CLINICAL TRIAL: NCT04810715
Title: Frequency of Pes Planus and Posterior Tibial Tendon Dysfunction in Patients With Ankylosing Spondylitis Ultrasonographic Study
Brief Title: Frequency of Pes Planus and Posterior Tibial Tendon Dysfunction in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: NEAS2021
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Posterior Tibial Tendon Dysfunction; Pes Planus; Spondylitis, Ankylosing
Keywords: Posterior Tibial Tendon Dysfunction; Ultrasonographic Evaluation; Pes Planus
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction; Flatfoot; Spondylitis, Ankylosing | interventions — HLA-B Antigens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: Anklyosing Spondilitis
  Interventions: Other: Patients with Ankylosing Spondylitis

INTERVENTIONS:
Other: Patients with Ankylosing Spondylitis — Observational study, not applicable

SUMMARY:
This investigation aims to investigate the frequency of pes planus and posterior tibial tendon dysfunction in patients with ankylosing spondylitis.

DETAILED DESCRIPTION:
Posterior tibial tendon dysfunction is the most common cause of acquired pes planus deformity in healthy adults. The posterior tibial tendon stabilizes the hindfoot against valgus and eversion forces and acts as a support along the medial longitudinal arch. If the posterior tibial tendon loses its functionality, the other ligaments of the foot and the joint capsule gradually weaken as the height of the medial longitudinal arch decreases or disappears, and it develops with pes planus. The presence of pes planus and spondyloarthropathy are also risk factors for the development of posterior tibial tendon dysfunction.

100 participants aged between 20-70 years with ankylosing spondylitis were planned to be included in this investigation. Posterior tibial tendon dysfunction frequency of patients with ankylosing spondylitis will be evaluated by both clinical examination and musculoskeletal ultrasonography device. The posterior tibial tendon will be evaluated by ultrasonography in terms of tendon diameter and fluid presence in 2 different locations in the retromalleolar area.

Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Ankylosing Spondylitis Quality of Life (ASQoL) Scale, Functional reach test, Timed up and go test, Berg Balance Scale, Dynamic and static balance with the Sportkat device will be used as evaluation parameters. It was planned that the evaluations were made once.

ELIGIBILITY:
Inclusion Criteria:

* Participitans who apply to the rheumatology outpatient clinic between the ages of 20-70 and who have been diagnosed with ankylosing spondylitis according to the Modified Newyork criteria will be included in this study.

  1. Ankylosing Spondilitis

Exclusion Criteria:

1. Malignity
2. Previous ankle surgery history
3. Muscle disease
4. Neuropsychiatric illnesses
5. İmbalance
6. Visual problems
7. Deafness

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Will be done only once on the first day after inclusion
  BASDAI includes six questions evaluating five important findings of the disease (Fatigue, hip and spine pain, swelling and pain in peripheral joints, enthesitis, duration and severity of morning stiffness). The pain levels of the patients will be evaluated with a Visual Analog scale (0: I have no pain, 10: I have very severe pain).
  Higher scores mean active disease.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Will be done only once on the first day after inclusion
  BASFI; consists of eight questions that evaluate the function of patients with AS and two questions that evaluate their daily life. Higher scores indicate greater limitations.
Ankylosing Spondylitis Quality of Life Scale (ASQOL) | Will be done only once on the first day after inclusion
  Ankylosing Spondylitis Quality of Life (ASQoL) scale is a disease-specific assessment parameter designed to measure health-related quality of life. It includes yes or no questions with a total score ranging from 0 to 18. The lower scores represent better quality of life.

SECONDARY OUTCOMES:
Functional reach test | Will be done only once on the first day after inclusion
  Functional reach test: It is the maximum distance that the participants can reach forward in the horizontal plane while maintaining her/his stability on the support surface in the standing position.
Timed up and go test (TUG) | Will be done only once on the first day after inclusion
  The TUG test is a simple evaluative test used to measure functional mobility. It uses the time that participants take to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. During the test, the participant is expected to wear their regular footwear and use any mobility aids that they would normally require.11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the worse scores.
Berg Balance Scale | Will be done only once on the first day after inclusion
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. The total score is 56. A score of < 45 indicates participants may be at greater risk of falling.
Foot and Ankle Outcome Score (FAOS) | Will be done only once on the first day after inclusion
  The FAOS is a 42-item questionnaire assessing patient-relevant outcomes in five separate subscales (Pain, other Symptoms, Activities of daily living, Sport and recreation function, foot and ankle-related Quality of life). Scores range from 0 to 100 with a score of 0 indicating the worst possible foot/ankle symptoms and 100 indicating no foot/ankle symptoms. Lower scores mean the worse scores.
Ultrasonographic evaluation of the posterior tibial tendon | Will be done only once on the first day after inclusion
  Posterior tibial tendon evaluation will be evaluated in 2 different locations in the retromalleolar area.Tendon diameter, continuity and fluid presence will be evaluated ultrasonographically. Power Doppler signal levels will be graded on a 4-point semi-quantitative scale (none-grade 0 / minor-grade 1 / middle-grade 2 / severe-grade 3).
Static and Dynamic Balance measurment with SportKAT Device. | Will be done only once on the first day after inclusion
  The SportKAT device used for determining postural oscillation consists of a balance platform and sensors that detect oscillations.There is a screen in front of the participant standing on the platform to provide feedback. During the static balance test, it is asked to keep the 'X' mark seen on the screen constant in the center. During the dynamic balance test, it is asked to to follow the moving cursor. The score range varies between 0 and 6000. The lower the score, the better the balance.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Arnoldner MA, Gruber M, Syre S, Kristen KH, Trnka HJ, Kainberger F, Bodner G. Imaging of posterior tibial tendon dysfunction--Comparison of high-resolution ultrasound and 3T MRI. Eur J Radiol. 2015 Sep;84(9):1777-81. doi: 10.1016/j.ejrad.2015.05.021. Epub 2015 May 21. PMID 26037267
- [Background] Guelfi M, Pantalone A, Mirapeix RM, Vanni D, Usuelli FG, Guelfi M, Salini V. Anatomy, pathophysiology and classification of posterior tibial tendon dysfunction. Eur Rev Med Pharmacol Sci. 2017 Jan;21(1):13-19. PMID 28121362
- [Background] Hasler P, Hintermann B, Meier M. Posterior tibial tendon dysfunction and MR imaging in rheumatoid arthritis. Rheumatol Int. 2002 May;22(1):38-40. doi: 10.1007/s00296-002-0183-1. PMID 12120910